CLINICAL TRIAL: NCT07252778
Title: Effect of a Short-term Multi-strain Probiotic Supplementation on the Exercise- Associated Gastrointestinal Disturbances in Trained Female Athletes Under Controlled Conditions During Professional Training Cycle
Brief Title: Effect of a Short-term Multi-strain Probiotic Supplementation in Endurance Athletes
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Krzysztof Durkalec-Michalski (Other)
Collaborators: Institute of Human Genetics, Polish Academy of Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Krzysztof Durkalec-Michalski, Prof., Poznan University of Physical Education
Organization: Poznan University of Physical Education (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZDS2025_0002
Record Dates: First submitted 2025-09-27; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Sports Nutrition; Biochemical Markers; Exercise Performance; Aerobic Capacity; Supplementation
Keywords: Probiotics; Gastro-intestinal markers; Microbiota; Rowing; Females

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPRO supplementation (Experimental): The experimental procedure for each participant in this group will include a 2-week period of MPRO supplementation.
  The entire study protocol will include familiarization and 4 main study visits (T1-T4; before/after supplementation). Enrolled volunteers will be randomly assigned to the treatment order with specific codes by an impartial biostatistician. Each study visit will consist of anthropometric indices and body composition evaluation, three saliva and blood samplings (resting; 3 min and 60 min after exercise) and exercise performance evaluation. Additionally, all participants will donate their stool samples into specially prepared two empty tubes. Samples will be collected on the same days as saliva/blood samples, early in the morning. Moreover, during each study visit, participants will complete a specific, validated GI symptoms questionnaire and specific and validated stress and mood questionnaires to assess their stress and mood before and after MPRO supplementation.
  Interventions: Dietary Supplement: MPRO supplementation
- PLA treatment (Placebo Comparator): The experimental procedure for each participant in this group will include a 2-week period of placebo supplementation.
  The entire study protocol will include familiarization and 4 main study visits (T1-T4; before/after supplementation). Enrolled volunteers will be randomly assigned to the treatment order with specific codes by an impartial biostatistician. Each study visit will consist of anthropometric indices and body composition evaluation, three saliva and blood samplings (resting; 3 min and 60 min after exercise) and exercise performance evaluation. Additionally, all participants will donate their stool samples into specially prepared two empty tubes. Samples will be collected on the same days as saliva/blood samples, early in the morning. Moreover, during each study visit, participants will complete a specific, validated GI symptoms questionnaire and specific and validated stress and mood questionnaires to assess their stress and mood before and after placebo supplementation.
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: MPRO supplementation — In the experimental procedure each athlete will be supplemented with a certificated, commercially available MPRO supplement SANPROBI® Barrier (Bifidobacterium lactis W52, Lactobacillus brevis W63, Lactobacillus casei W56, Lactococcus lactis W19, Lactococcus lactis W58, Lactobacillus acidophilus W37, Bifidobacterium bifidum W23, Bifidobacterium lactis W51, Lactobacillus salivarius W24).
  The supplement will be provided in the capsule form and will be taken twice a day [4 capsules of MPRO/day (2×10to9 CFU/g, 500 milions CFU/capsule) in two servings/day (2x2 capsules].
  Arms: MPRO supplementation
Dietary Supplement: Placebo treatment — In the control procedure each athlete will be supplemented with a placebo (PLA). The PLA group will receive corn starch mixed with maltodextrins. The PLA will be provided in the capsule form and will be taken twice a day (2x2 capsules/day).
  Arms: PLA treatment

SUMMARY:
The aim of this project is to evaluate and identify the effect of a short-term 2-week multi-strain probiotic (MPRO) supplementation on the exercise-associated gastrointestinal (GI) symptoms and perturbations in high level female athletes of the Polish national team during strictly controlled conditions of a training camp, based on recommendations for best practices for probiotic (PRO) research in athletes and assessment of EX-associated GI perturbations.

DETAILED DESCRIPTION:
Objective of the study: GI health is crucial for the maintenance of general health and high performance in athletes. It is well known that GI symptoms are common in endurance athletes and that women are more likely to experience moderate or severe levels of symptoms. Exercise stress and external factors have an impact on GI health, leading to perturbations of GI integrity and functions negatively affecting performance outcomes. It is therefore necessary to develop treatment strategies capable of strengthening the GI health. Among the various preparations, PRO seem to induce improvements in intestinal diseases. There is a possible direct association between the reduced exercise-induced perturbations and cytokines, gut barrier function, and GI symptoms after PRO supplementation, but it has not been fully clarified yet. Moreover, it is stated that PRO benefits are strain-specific and dose-dependent, and include improved gut-barrier function, nutrient absorption, recovery and performance in athletes. Nevertheless, there is lack of well-designed studies on athletes population. Therefore, the main goal of the project is to evaluate and identify the effect of a short-term 2-week MPRO supplementation on the exercise- associated GI symptoms and perturbations in high level female rowers (particularly exposed to GI disturbances) of the Polish national team during completely controlled conditions of a training camp, based on recommendations for best practices for probiotic research in athletes and assessment of exercise-associated GI perturbations. The primary outcome is to recognize the MPRO supplementation effect on GI mechanisms, responsible for the occurrence of exercise-induced GI symptoms negatively affecting exercise performance. The following research hypotheses were adopted: A) considerable physical stress induced by high intensity exercises during national training camp contribute to the occurrence of GI disturbances; B) MPRO during high intensity training schedule may have a significant impact on specific key markers of GI perturbations; C) MPRO may have a positive effect on GI integrity; D) MPRO may have a beneficial effect on the systemic immune responses; E) MPRO may alter the fecal bacterial composition; F) MPRO may positively affect psychological stress and mood during high intensity training camp; G) MPRO may positively affect exercise performance outcomes.

Research project methodology: The study will be conducted in the standard of randomized, triple-blind, PLA-controlled crossover studies. A number of 30 high level female rowers will be enrolled. Specific MPRO strategy will be implemented. The assessment of body composition, exercise performance, baseline stool and baseline/post-exercise blood collection, GI and stress and mood status and nutrition will be performed. Samples will be analysed for: A) GI integrity markers permeability, bacterial endotoxin translocation, B) immune/stress responses' markers [inflammatory cytokine profile, immune cell response, C) exercise adaptation and intensity markers, D) stool GI integrity markers, E) fecal bacterial composition.

Expected impact of the research project on the development of science, practice and society: This completely innovative MPRO project will be conducted according to recently released recommendations for best practices for probiotic research in athletes and assessment of exercise-associated GI perturbations. Furthermore, recognizing the impact of MPRO on GI health could have beneficial implications for athletes, and people from the general population. An indisputable strength of our project is the fact that obtained data may be extrapolated into a real-world. Information on whether MPRO administration promotes proper GI health and physical training adaptation could be important for developing recommendations for PRO usage. Finally, the indisputable necessity of conducting research in the area of PRO is proved, in particular, by the abundance of GI disturbances, in terms of investigating natural methods in the prevention of GI symptoms.

ELIGIBILITY:
Inclusion Criteria:

* belonging to the national rowing team;
* training experience ≥5 years;
* a currently issued medical certificate confirming
* good health and capacity to practice sports;
* good health without chronic health disorders;
* written informed consent to participate.

Exclusion Criteria:

* injury, any health contraindication or failure to perform exercise procedures;
* gastrointestinal infections, diseases, disorders;
* past history of gastrointestinal surgery, and
* other self-reported gastrointestinal issues;
* reporting symptoms of infection or taking any medication (e.g. antibiotics) for 4 weeks before the study protocol;
* current supplementation of prebiotics,
* probiotics, synbiotics (last 4 weeks);
* current intake of pharmaceutical agents (e.g., nonsteroidal anti-inflammatory drugs, laxatives, antidiarrhea agents, antacids, and/or antiemetics) (last 4 weeks);
* failure to follow the study protocol;
* declared general feeling of being unwell;
* pregnancy or current pregnancy planning.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in gastrointestinal integrity and inflammation markers (I-FABP, claudin-3, zonulin, LPS, scd-14, LBP, ocludin, lipocalin-2, DAO) (ng/mL) in blood after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the gastrointestinal integrity markers (I-FABP, claudin-3, zonulin, LPS, scd-14, LBP, ocludin, lipocalin-2, DAO) (ng/mL) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in gastrointestinal integrity and inflammation markers (zonulin, ocludin, lipocalin-2) (ng/mL) in stool after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the gastrointestinal integrity markers (zonulin, ocludin, lipocalin-2) (ng/mL) in stool at rest will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in gastrointestinal integrity and inflammation markers (calprotectin, lactoferrin) (μg/g) in stool after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the gastrointestinal integrity markers (calprotectin, lactoferrin) (μg/g) in stool at rest will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in gastrointestinal integrity and inflammation markers (α-1 antitripsin) (mg/g) in stool after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the gastrointestinal integrity markers (α-1 antitripsin) (mg/g) in stool at rest will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in gut microbiota phylogenetic diversity (Faith's phylogenetic diversity index) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of phylogenetic α-diversity of the gut microbiome assessed from stool 16S rRNA gene sequencing; computed as Faith's Phylogenetic Diversity (sum of branch lengths on the phylogenetic tree corresponding to observed taxa) at rest will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in gut microbiota species diversity (Shannon diversity index) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of species (taxonomic) α-diversity of the gut microbiome assessed from stool 16S rRNA gene sequencing; computed using the Shannon diversity index (accounts for richness and evenness) at rest will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in gut microbiota species richness (number of observed species (OTUs)) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of species richness of the gut microbiome assessed from stool 16S rRNA gene sequencing; reported as the number of observed operational taxonomic units (Observed OTUs) at rest will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).

SECONDARY OUTCOMES:
Changes in blood cytokines (IL-1β/1ra/6/8/10/17, TNF-α) (pg/mL) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the cytokines (IL-1β/1ra/6/8/10/17, TNF-α) (pg/mL) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in stress marker (cortisol) (ng/ml) in blood and saliva after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the stress marker (cortisol) (ng/ml) in blood and saliva at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in saliva SIgA concentration (μg/mL) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the saliva SIgA concentration (μg/mL) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in gastrointestinal symptoms incidence and severity (points) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the gastrointestinal symptoms incidence and severity (points) will be carried out before, during and after aerobic fitness and exercise performance test at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in psychological stress and mood (points) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the psychological stress and mood (points) will be carried out at rest at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in white blood cells count and differential (count/L) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the leukocytes (neutrophils, monocytes, lymphocytes, neutrophils:lymphocytes ratio) (count/L) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in white blood cells count and differential (%) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the leukocytes (neutrophils, monocytes, lymphocytes, neutrophils:lymphocytes ratio) (%) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA)

OTHER OUTCOMES:
Changes in the aerobic fitness and exercise performance test results (aerobic capacity measured by maximum workload at exhaustion in Watts) after MPRO supplementation and PLA treatment IRT performance | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the aerobic capacity (Watts) will be carried out by the increasing intensity ramp exercise test on a rowing ergometer at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in the aerobic fitness and exercise performance test results (aerobic capacity measured by maximal oxygen uptake in mL/min/kg) after MPRO supplementation and PLA treatment IRT performance | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the aerobic capacity (maximal oxygen uptake in mL/min/kg) will be carried out by the increasing intensity ramp exercise test on a rowing ergometer at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in heart rate (bpm) during aerobic fitness and exercise performance test after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the heart rate (bpm) during the increasing intensity ramp exercise test on a rowing ergometer will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in lactate concentration (mmol/L) before, during and after aerobic fitness and exercise performance test after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the lactate concentration (mmol/L) will be performed from fingertip capillary blood before, during and 3-min after the increasing intensity ramp exercise test on a rowing ergometer at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in glucose concentration (mg/dL) before, during and after aerobic fitness and exercise performance test after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the glucose concentration (mmol/L) will be performed from fingertip capillary blood before, during and 3-min after the increasing intensity ramp exercise test on a rowing ergometer at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in gasometry markers (pH) before, during and after aerobic fitness and exercise performance test after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the gasometry markers (pH) will be performed from fingertip capillary blood before, during and 3-min after the increasing intensity ramp exercise test on a rowing ergometer at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in gasometry markers (pCO2, pO2) (mmHg) before, during and after aerobic fitness and exercise performance test after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the gasometry markers (pCO2, pO2) (mmHg) will be performed from fingertip capillary blood before, during and 3-min after the increasing intensity ramp exercise test on a rowing ergometer at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in electrolites' concentration (Ca, Na, K, Cl) (mmol/L) before, during and after aerobic fitness and exercise performance test after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the electrolites' concentration (Ca, Na, K, Cl) (mmol/L) will be performed from fingertip capillary blood before, during and 3-min after the increasing intensity ramp exercise test on a rowing ergometer at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in nutritional status indices (concentration of total protein and albumin) (g/dL) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the nutritional status indices (concentration of total protein and albumin) (g/dL) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in nutritional status indices (concentration of urea) (mmol/L) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the nutritional status indices (concentration of urea) (mmol/L) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in muscle damage markers (concentration of creatinine) (μmol/L) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the muscle damage markers (concentration of creatinine) (μmol/L) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in muscle damage markers (activity of alanine aminotransferase, aspartate aminotransferase, creatine kinase, lactate dehydrogenase) (U/L) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the muscle damage markers (activity of alanine aminotransferase, aspartate aminotransferase, creatine kinase, lactate dehydrogenase) (U/L) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in hematological indices (red blood cells, RBC) (count/L) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the hematological indices (red blood cells, RBC) (count/L) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in hematological indices (hemoglobin concentration, HGB) (mmol/L) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the hematological indices (hemoglobin concentration, HGB) (mmol/L) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in hematological indices (hematocrit, HCT) (L/L) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the hematological indices (hematocrit, HCT) (L/L) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in hematological indices (mean corpuscular volume, MCV; mean platelet volume, MPV) (fL) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the hematological indices (mean corpuscular volume, MCV; mean platelet volume, MPV) (fL) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in hematological indices (mean corpuscular hemoglobin mass, MCH) (fmol) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the hematological indices (mean corpuscular hemoglobin mass, MCH) (fmol) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in hematological indices (mean corpuscular hemoglobin concentration, MCHC) (mmol/L) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the hematological indices (mean corpuscular hemoglobin concentration, MCHC) (mmol/L) after at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in hematological indices (platelet count, PLT) (count/L) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the hematological indices (platelet count, PLT) (count/L) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in hematological indices (platelet hematocrit, PCT) (cL/L) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the hematological indices (platelet hematocrit, PCT) (cL/L) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in hematological indices (platelet distribution width, PDW; platelet large cell ratio, PLCR; red blood cells distribution width - coefficient of variation, RDW-C) (%) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the hematological indices (platelet distribution width, PDW; platelet large cell ratio, PLCR; red blood cells distribution width - coefficient of variation, RDW-C) (%) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Changes in hematological indices (red blood cells distribution width - standard deviation, RDW-S) (fL) after MPRO supplementation and PLA treatment | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of the hematological indices (red blood cells distribution width - standard deviation, RDW-S) (fL) after at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the test exercise [REC]) will be carried out at four main visits to the laboratory (T1-T4; before/after supplementation with MPRO and PLA).
Analysis of body composition (fat-free mass, fat mass) (kg) | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of body composition (fat-free mass, fat mass) (kg) will be carried out before the execution of exercise protoMPROs on each research visit.
Analysis of body composition (fat-free mass, fat mass) (%) | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of body composition (fat-free mass, fat mass) (%) will be carried out before the execution of exercise protoMPROs on each research visit.
Analysis of body composition (total body water) (L) | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of body composition (total body water) (L) will be carried out before the execution of exercise protoMPROs on each research visit.
Analysis of body composition (total body water) (%) | Baseline (before MPRO supplementation) and after 2 weeks of MPRO supplementation; baseline (before PLA supplementation) and after 2 weeks of PLA supplementation.
  Assessment of body composition (total body water) (%) will be carried out before the execution of exercise protoMPROs on each research visit.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Durkalec-Michalski, PhD, Study Chair — Department of Sports Dietetics, Poznan University of Physical Education Poznań
Locations (1):
- Department of Sports Dietetics, Poznan University of Physical Education Poznań, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
Shared data will be exclusively related to the level of recorded indicators, without personal data. The data obtained will be attached to scientific publications, depending on the requirements of the journal.
  De-identified individual participant data (IPD), including timepoint-specific values of primary and secondary outcome measures (e.g., performance results, hematological and physiological parameters), will be shared. Data will be made available upon reasonable request to qualified researchers for non-commercial academic purposes, following publication of the primary results. Requests should be directed to the corresponding author via institutional email. A data use agreement may be required.